CLINICAL TRIAL: NCT06309004
Title: Development, Feasibility, Efficacy, and Cost-effectiveness of an Online ACT Intervention for Disorders of Gut-Brain Interaction (Sub-study 1)
Brief Title: Development of an Online ACT Intervention for Disorders of Gut-Brain Interaction
Acronym: iACTforDGBI
Status: Active, not recruiting | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: Uppsala University (Other); SahlgrenskaUniversityHospital (Unknown); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00741a
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anxiety and Depression; Disorders of Gut-brain Interaction
Keywords: DGBI; ACT; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults with DGBI: Adults with DGBI, and clinically meaningful symptom levels of anxiety and/or depression
- Healthcare professionals: Healthcare professionals (physicians, psychologists, nurses, and dietitians).

SUMMARY:
The goal of this clinical trial is to develop and test the iACTforDGBI intervention in a sample of Swedish individuals with DGBI (Disorders of Gut-Brain Interaction).

The first substudy of this project (Substudy 1) aims to answer the following question: How can the design of iACTforDGBI be tailored to meet the specific needs of individuals with DGBI and clinically meaningful symptoms of anxiety and depression?

Participants (individuals with symptoms compatible with a DGBI and anxiety and/or depression, and healthcare professionals working with DGBI patients) will be asked to participate in online focus-group interviews and provide information on their views of a preliminary version of the iACTforDGBi intervention.

ELIGIBILITY:
DGBI participants:

Inclusion Criteria:

1. Age between 18 and 75 years;
2. Exhibiting clinical symptom severity for at least one DGBI diagnosis (assessed with the Rome IV Diagnostic Questionnaire for Functional Gastrointestinal Disorders in Adults (Palsson et al., 2016));
3. Clinically meaningful levels of depressive symptoms or anxiety: score ≥ 13 on the Montgomery Åsberg Depression Rating Scale (MADRS; depressive symptoms), or score ≥ 10 on the Generalized Anxiety Disorder scale-7 (GAD-7; anxiety symptoms; Spitzer et al., 2006);
4. Stable medication for psychiatric symptoms including anxiety, depression, and sleep problems for at least two months prior to intervention;
5. Ability to read and write Swedish;
6. Access to a device (like a computer, tablet, or smartphone) with access to the internet and that can be used to attend video conferences and preview the intervention platform (i.e., have a microphone and speakers or headphones).

Exclusion Criteria:

1. Currently undergoing any form of psychological intervention;
2. Increased risk of suicide (≥4 points on MADRS item 9);
3. Severe depression (≥34 points on MADRS).

Healthcare professionals:

Inclusion Criteria:

a) Being a healthcare professional currently working with DGBI patients and/or with ACT-based/digital interventions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with DGBI:
  People with clinically meaningful symptom severity of DGBI, and depression and/or anxiety.
  Healthcare professionals:
  Physicians, psychologists, nurses, and dietitians working from different regions in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Focus group interviews | 60-90 minutes per interview
  Focus group interviews

CONTACTS AND LOCATIONS:
Overall Officials: Inês A Trindade, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This question is under investigation. Some of our data contain sensitive information on health, and the main priority is participants integrity which need to be balanced against basic scientific principles on scrutiny. However, any personal data that can be shared without compromising participants integrity to a reasonable degree will be shared upon reasonable request.